CLINICAL TRIAL: NCT06649838
Title: Customized Circulating Tumor DNA Testing for Cervical Cancer Recurrence Surveillance and Treatment Decisions
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RCC-ctDNA
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-10

CONDITIONS: Immunotherapy; Cervical Cancer; CtDNA; Biomarker
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Immunotherapy is the main option for advanced, recurrent and metastatic cervical cancer. However, due to the complex interaction between the immune system and tumors, there is still a lack of effective markers for immunotherapy. Scientists are actively searching for and developing new immunotherapy markers. For cervical cancer diagnosis, it has been shown that ctDNA mutations can reflect HPV integration sites. In terms of cervical cancer prognosis monitoring, cohort studies focused on the application of HPV ctDNA in the field of cervical cancer prognosis monitoring. The aim of this study is to design a customized ctDNA probe for cancer patients through a priori tumor detection method, and to guide recurrence monitoring plan and implement individualized adjuvant therapy according to the results, and to explore personalized biomarkers to guide cervical cancer immunotherapy. To explore the possibility of customized ctDNA detection as a diagnostic marker for cervical cancer. To explore the predictive and prognostic value of customized ctDNA dynamic monitoring. A multi-arm cohort clinical study is planned. To comprehensively study the treatment strategy of advanced and recurrent cervical cancer and explore the related biomarkers through the customized dynamic monitoring of ctDNA in patients with advanced and recurrent cervical cancer. A total of 60 patients with cervical cancer were enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. be willing and able to provide written informed consent/consent for the trial.
2. Be 18 years of age or older on the date of signing the informed consent form.
3. patients with histologically or cytologically documented locally advanced, advanced, or first recurrent cervical cancer. For treatment-naive patients, 4) no previous cancer treatment including chemotherapy or radiotherapy; Patients with an initial recurrence had not received any other cancer treatment, including chemotherapy or radiotherapy, after the diagnosis of an initial recurrence before enrollment.

5) measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

6) willing and able to provide tumor lesions or excisional biopsy tissue. 7) a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale. Demonstrate adequate organ function.

8) a negative pregnancy test in a fertile female patient.

Exclusion Criteria:

1. be diagnosed as immunocompromised or receiving systemic steroid therapy or any other form of immunosuppressive therapy.
2. a known history of active tuberculosis (Mycobacterium tuberculosis).
3. have a known other malignancy that is progressing or requires active treatment.
4. known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
5. have an active autoimmune disease requiring systemic treatment within the past 2 years.
6. known history or any evidence of active noninfectious pneumonia.
7. active infection requiring systemic therapy.
8. there is historical or current evidence of any condition, treatment, or laboratory abnormality that could confound the trial results, interfere with the patient's participation throughout the trial, or that the treatment investigator believes participation would not be in the patient's best interest.
9. psychiatric or substance abuse disorders known to interfere with compliance with trial requirements.
10. be pregnant or breastfeeding, or expect to become pregnant or give birth to a child within the intended duration of the trial.
11. had a known history of human immunovirus (HIV) (HIV 1/2 antibodies).
12. known to have active hepatitis B (e.g., HBsAg reactive) or hepatitis C.
13. received live vaccine within 30 days of planned initiation of study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 60 patients with cervical cancer were enrolled, including 10 patients with local advanced cervical cancer (IB3-IIB) and 20 patients with advanced cervical cancer (10 patients with stage IIIC and 10 patients with stage IV). The second team consisted of 30 patients with recurrent cervical cancer.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-03-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Somatic mutation detection by WES | from Des 2024 to Oct 2026